CLINICAL TRIAL: NCT02798172
Title: The Effect of Alogliptin on Pulmonary Function in Obese Patients With Type 2 Diabetes Inadequately Controlled by Metformin Monotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fourth People's Hospital of Shenyang (Other)
Responsible Party: Principal Investigator, Jin-song Kuang, Chief physician, Fourth People's Hospital of Shenyang
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20140508
Record Dates: First submitted 2016-05-30; First posted 2016-06-14 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2016-06

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — alogliptin; Metformin

ARMS (2):
- Alogliptin+metformin (Experimental): Alogliptin (alogliptin benzoate) is the most recent DPP-4 inhibitor; it entered the market in 2006. It is a potent and highly selective DPP-4 inhibitor with oral antidiabetic activity; Metformin is the most commonly prescribed first-line drug worldwide for the treatment of T2DM, it acts by decreasing both hepatic glucose production and intestinal glucose absorption, while improving insulin sensitivity, metformin as a safe and valid oral antidiabetic drug was recommended to the obese patients with a body mass index (BMI) >30 kg/m2, it has some value in reducing or preventing weight gain and changes in metabolic parameters during treatment, and it can be combinated with other antidiabetic drug
  Interventions: Drug: Alogliptin and Metformin
- metformin (Experimental): Metformin is the most commonly prescribed first-line drug worldwide for the treatment of T2DM, it acts by decreasing both hepatic glucose production and intestinal glucose absorption, while improving insulin sensitivity, metformin as a safe and valid oral antidiabetic drug was recommended to the obese patients with a body mass index (BMI) >30 kg/m2, it has some value in reducing or preventing weight gain and changes in metabolic parameters during treatment, and it can be combinated with other antidiabetic drug
  Interventions: Drug: Alogliptin and Metformin

INTERVENTIONS:
Drug: Alogliptin and Metformin — The patients in the control group were given metformin (1,000 mg, bid po) and the patients in the intervention group were given metformin (500 mg, bid po) combined with alogliptin (25 mg, qd po)

SUMMARY:
Objective: To observe the effect of alogliptin combined with metformin on pulmonary function in obese patients with type 2 diabetes inadequately controlled by metformin monotherapy (500 mg, bid po, for at least 3 months), and evaluate its efficacy and safety.

Method: After a 2-week screening period, adult patients (aged 36-72 years) entered a 4-week run-in/stabilization period. Then, patients were randomly assigned to either the intervention group (n=55) or control group (n=50) for 26 weeks. The patients in the control group were given metformin (1,000 mg, bid po) and the patients in the intervention group were given metformin (500 mg, bid po) combined with alogliptin (25 mg, qd po). All the patients received counseling about diet and exercise from a nutritionist during run-in and treatment periods.

The primary endpoints were the between-group differences in the changes pulmonary function parameters [VC%, FVC%, FEV1%, PEF%, MVV%, TLC%, FEV1/FVC%, DLCO%, and DLCO/VA%] between pretherapy and posttreatment. The secondary endpoints were changes from baseline to week 26 in HbA1c, FPG, 2hPG, HOMA-IR, WC, and BMI. The tertiary endpoints were the changes from baseline to week 26 in blood-fat (TC, HDL-C, LDL-C, and TG). The quartus endpoints were the changes from baseline to week 26 in SBP and DBP. The fifth endpoints were the changes from baseline to week 26 in oxidative/antioxidative parameters (ROS, MDA, SOD, and GSH-PX). In addition, safety endpoints were assessed (AEs, clinical laboratory tests, vital signs, and electrocardiographic readings).

DETAILED DESCRIPTION:
Alogliptin was provided by Takeda Chemical industries Ltd in Japan, trade name: Nesina, 25 mg/tablet. Metformin was provided by Bristol Myers Squibb in America, trade name: Glucophage, 500 mg/tablet. Research kits for ROS, MDA, and SOD, GSH-PX were provided by Nanjing Jiancheng Bioengineering Institute in China. Research kits for TC, HDL-C, HDL-C, and TG were provided by were provided by Nanjing Jiancheng Bioengineering Institute in China. The spirometer used for pulmonary function tests was provided by Jaska Corporation in Japan, model number: HI-101

ELIGIBILITY:
Inclusion Criteria:

* 1) Aged from 36 to 72 years of either gender; 2) BMI >28.0 kg/m2, and WC >90 cm (male), or WC >85 cm (female); 3) The patients were diagnosed with T2DM and the serological outcome (7.0%<HbA1c<10.0%) did not reach the therapeutic targets and oral metformin monotherapy (500 mg, bid po, ≥3 months prior to screening); 4) No smoking history, pulmonary disease nor pulmonary infection within a fortnight; 5) Did not have hepatopathy, nephropathy and gastrointestinal disease; and 6) Likely to have good compliance and able to visit our hospital for periodic assessments.

Exclusion Criteria:1) T1DM, gestation and lactation; 2) Renal inadequacy; 3) hypohepatia; 4) Intensive care with insulin treatment; 5) Intolerance to alogliptin and metformin; 6) Heart failure; 7) Had received antidiabetic agents; 8) Antihypertensive drugs can not control the BP adequately or severe uncontrolled hypertension; 9) Cholesterol-lowering drugs can not control the blood-fat adequately; and 10) Use of weight loss drugs.

-

Ages: 36 Years to 72 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2014-05; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
The primary endpoints were changes from baseline to week 26 in pulmonary function parameters [VC%, FVC%, FEV1%, PEF%, MVV%, TLC%, FEV1/FVC%, DLCO%, and DLCO/VA%] between pretherapy and posttreatment. | 26 weeks

SECONDARY OUTCOMES:
The secondary endpoints were changes from baseline to week 26 in HbA1c in intervention group (n=44) and control group (n=37). | 26 weeks
The tertiary endpoints were the changes from baseline to week 26 in blood-fat (TC, HDL-C, LDL-C, and TG) in the intervention group (n=44) and control group (n=37). | 26 weeks
The fourth endpoints were the changes from baseline to week 26 in FPG, 2hPG in the intervention group (n=44) and control group (n=37). | 26 weeks
The fourth endpoints were the changes from baseline to week 26 in oxidative/antioxidative parameters (ROS, MDA, SOD, and GSH-PX) in the intervention group (n=44) and control group (n=37). | 26 weeks
In addition, safety endpoints were assessed (AEs, clinical laboratory tests, vital signs, and electrocardiographic readings) | 26 weeks

OTHER OUTCOMES:
The changes of BMI from baseline to week 26 in intervention group (n=44) and control group (n=37). | 26 weeks